CLINICAL TRIAL: NCT06531330
Title: Use of Tools for Early Detection of Cerebral Palsy: A Study on Pediatric Physiotherapists in Turkey
Brief Title: Use of Tools for Early Detection of Cerebral Palsy
Acronym: tooluse
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Collaborators: Gazi University (Other); Karadeniz Technical University (Other); Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Asistant Professor, Kahramanmaras Sutcu Imam University
Other Study IDs: KahramanmarasSIU2
Record Dates: First submitted 2024-07-24; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Palsy; Early Developmental Impairment; Infant Development
Keywords: Cerebral Palsy; Early Detection; tools; Pediatric Physiotherapists
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Pediatric physiotherapists working in Turkey

SUMMARY:
High risk of infant is defined as an infant who has a history of negative environmental and biological factors and these factors can cause neuromotor development problems. This group is a heterogeneous group that includes premature babies born under thirty-seven weeks, term babies with low birth weight (LBW), or babies with developmental delays for various reasons. These infants are also monitored for Cerebral Palsy (CP). CP is the most common physical disability in childhood, with an incidence of 2.1 per 1000 births.In a 2017 clinical review of early diagnosis tools, a group of international experts published best practice recommendations, calling for early diagnosis to be made as a result of timely use of the recommended tools. The diagnosis of CP is typically made by a physician between 12 and 24 months of age, but in some cases it is delayed until 42 months.Correct and early use of the key tools required for early diagnosis may allow much earlier detection of CP for infants younger than 5 months or older.Early detection and monitoring of infants in the community for CP is essential only with appropriate, valid and reliable tools in order to minimize possible sequelae through timely implementation of CP-specific interventions. According to international guidelines, babies with high risk of CP should be followed up. This follow-up should be done by an interdisciplinary team such as neonatologist, pediatrician, pediatric neurologist, physiotherapist, speech-language-swallowing therapist, and special education specialist. Pediatric physiotherapists are an important part of this team in terms of developmental follow-up and rehabilitation. Therefore, it is important that the awareness level of pediatric physiotherapists in this field in our country is sufficient, they are equipped with various trainings and reach the international level. In this way, families at risk of CP can provide early guidance for their children, ensure early diagnosis of CP, and initiate treatment.The aim of this study is to evaluate the use of early diagnostic evaluation tools in at-risk of infants between the ages of 0-2 at risk of CP in pediatric physiotherapy practice in Turkey.

DETAILED DESCRIPTION:
Prematures make up the majority of risky babies; perinatal asphyxia, hypoxic ischemic encephalopathy (HIE), periventricular leukomalacia (PVL), intraventricular hemorrhage (IVH), respiratory distress syndrome (RSD), bronchopulmonary dysplasia (BPD), hyperbilirubinemia, viral infections, fetal alcohol syndrome, muscle tone disorders, hydrocephalus and They may encounter risk factors such as microcephaly.It is important to detect early atypical neurodevelopmental findings that may occur in at-risk of infants at later ages and direct them to the necessary intervention programs.In this context, all healthcare professionals in the follow-up of at-risk babies should follow developmental and medical follow-up guidelines and use various neuromotor assessment methods. It is also stated in the guidelines of the American Academy of Pediatrics (APA) and the high-risk baby monitoring guide of the Turkish Neonatology Association that these babies should be monitored periodically by a team.The importance of monitoring all premature infants, especially very low birth weight (VLBW) babies <1500g, at least twice in the first year of their lives, with age-appropriate neuromotor and developmental evaluations is emphasized. In this way, infants; By determining motor, sensory, cognitive and social developmental delays, developmental problems in later ages can be predicted. In addition, physiotherapy and rehabilitation or special education needs can be determined in terms of early intervention and motor development, and early referral to appropriate support programs can be provided.The 3 methods with the best predictable validity that can determine CP before the corrected 5-month period are; Neonatal MRI (86%-89% sensitivity), Prechtl's GMs Evaluation (98% sensitivity), HINE (90% sensitivity). Using the HINE test alone was also found to be reliable in determining the development of CP. In recent years, studies have shown that the diagnosis of high-risk CP can be detected at the 3rd month with predictive validity and reliability by evaluating the quality of Prechtl's GMs movements.Early physiotherapy and rehabilitation in CP includes approaches starting from the neonatal period and up to 24 months. The main aim is to provide normal functional movements and normal sensory input by using the rapid learning ability resulting from brain plasticity.Velde et al. In order to implement a new evidence-based clinical guideline for early diagnosis in Australia, a study aimed to determine the age at diagnosis, suitability for recommended tests, and acceptability of the early diagnosis clinic for parents and referrers, by following patients according to international guidelines, estimated CP diagnosis between 4-8 months. They showed. The follow-up clinic in this study was found to be highly acceptable to parents and referrers. During this follow-up period, pediatricians had the highest referral rates (39%), followed by auxiliary healthcare professionals (31%), primary caregivers (14%) and other healthcare professionals (16%).In a study conducted among American pediatricians, it was stated that there was uncertainty about how to diagnose and refer babies with motor delays, and variability in knowledge and practices regarding the identification of motor delays in these babies. A study conducted with clinicians (pediatricians, physiotherapists and occupational therapists) in New Zealand investigated current clinical practices regarding awareness and use of diagnostic tools for the detection of CP. Despite high awareness of the risk of CP in New Zealand, current use of international best practice tools in the clinic has been observed to be low. Clinicians who do not make diagnoses within their professional roles also reported that the assessment tools were rarely used, with 74% never using GMs or HINE and 54% in assessing children at risk for CP. Barriers to use have been cited as lack of time or funding, lack of clear guidelines, and inadequate management support. In a study conducted with pediatric physiotherapists in Spain, the average age at which CP was suspected was 12.6 months. To evaluate and diagnose the risk of CP, most physiotherapists; stated that they used the child's clinical history (88.1%), AIMS (41.3%) and Vojta Assessment Procedure (32.1%). In Spain, physiotherapists were found to rarely use GMs (25.7%) and HINE (28.4%). These results showed that pediatric physiotherapists in Spain rely on clinical history and older tools to identify children with CP.In this study, it was aimed to determine the awareness levels about the importance of the use of these tools in terms of early diagnosis and intervention in CP in Turkey, the frequency of use and the reasons for the obstacles if they cannot be used. In this context, the awareness levels of physiotherapists in Turkey will be determined through a digital survey administered digitally to pediatric physiotherapists in Spain and translated into Turkish after obtaining the necessary permissions.

ELIGIBILITY:
Inclusion Criteria:

- Physiotherapists who have been working in the field of pediatric physiotherapy for at least 3 years

Exclusion Criteria:

* Physiotherapists with any psychiatric diagnosis

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Physiotherapists who have been working in the field of pediatric physiotherapy for at least 3 years and aged between 25-50 years old will be included in the study.Physiotherapists with any psychiatric diagnosis will be excluded.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Digital survey | The baseline of the study for one time
  Digital survey: Purpose-developed digital survey consisting of 45 multiple choice questions with 5 thematic sections. The survey to be used in this context will be a survey administered digitally to pediatric physiotherapists in Spain and translated into Turkish after obtaining the necessary permissions. This survey will be administered via Google forms.Pediatric physiotherapists working in different clinics will be asked to fill out a purpose-built electronic survey online. All survey questions will be delivered to physiotherapists electronically via social media (Whatsapp, Instagram, Facebook) or e-mail. Pediatric physiotherapists from at least 20 different provinces in Turkey will participate in this study.
  The survey measure will be assessed at the baseline of the study for one time.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Adiguzel, PhD PT, Principal Investigator — Kahramanmaras Sutvu Imam University; Bulent Elbasan, Proffessor, Study Director — Gazi University
Locations (1):
- Hatice, Kahramanmaraş, Turkey (Türkiye)